CLINICAL TRIAL: NCT07160660
Title: Patients' Satisfaction and Clinical Investigation of Removable Partial Denture Anchorage With Extracoronal Adhesive Attachments in Comparison With Clasp-retained Partial Dentures
Status: Not yet recruiting | Type: Observational
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Florence Auderset, Member of Research Group of the Department of Clinical Research, Principal Investigator, Dr. med. dent., University of Basel
Other Study IDs: PSCI2025
Record Dates: First submitted 2025-08-24; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Extracoronal Adhesive Attachment; Clasp-retained Partial Dentures; Patients Satisfaction With Removable Dental Prostheses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with extracoronal adhesive attachments as retentive elements of RPD (group A): RDP = removable dental prostheses
  Interventions: Other: Patients' satisfaction and clinical investigation of removable partial denture anchorage with extracoronal adhesive attachments
- Patients with clasps as retentive elements of RPD (group B): RDP = removable dental prostheses
  Interventions: Other: Patients' satisfaction and clinical investigation of removable partial denture anchorage with conventional clasps

INTERVENTIONS:
Other: Patients' satisfaction and clinical investigation of removable partial denture anchorage with extracoronal adhesive attachments — * Completion of a questionnaire by the participant, including patient satisfaction on VAS (visual analogue scale) and prostheses usability, clinical examination of the remaining dentition, the abutment teeth of the extracoronal adhesive attachment and the RPD.
  * Evaluation of the attachment's condition, retention, and any signs of biological or technical complications.
  * Collection of relevant medical and dental history from patients' records (consent provided).
  Groups: Patients with extracoronal adhesive attachments as retentive elements of RPD (group A)
Other: Patients' satisfaction and clinical investigation of removable partial denture anchorage with conventional clasps — * Completion of a questionnaire by the participant, including patient satisfaction on VAS (visual analogue scale) and prostheses usability, clinical examination of the remaining dentition, the abutment teeth of the clasps and the RPD.
  * Evaluation of the clasps' condition, retention, and any signs of biological or technical complications.
  * Collection of relevant medical and dental history from patients' records (consent provided).
  Groups: Patients with clasps as retentive elements of RPD (group B)

SUMMARY:
Removable partial dentures (RPD) are a well-established treatment option for the prosthetic rehabilitation of partially edentulous patients. They are retained at the remaining natural teeth by clasps to provide functional stability. As an alternative to clasps extacoronal adhesive attachments are fixed to the abutment teeth using adhesive cementation techniques. These adhesive attachments improve retention and stability of the prostheses and are indicated when the patient requires a non-visible retention element and healthy coronal tooth structure is available as a prerequisite. In clinical practice, extracoronal adhesive attachments offer a minimally invasive and aesthetic anchoring alternative of removable dental prostheses associated with higher costs compared to a common clasp retention. As a result, adhesive attachments are relatively rarely used and are technically sensitive both in the clinical realisation and in terms of the dental technology. Hence, limited scientific data are available regarding their long-term clinical behaviour, but no data is available about patients' satisfaction with such extracoronal adhesive attachments.

This research project aims to investigate patients' satisfaction with extracoronal adhesive attachments (group A) of removable dental prostheses in comparison to clasps (group B), and to investigate the short- and long-term clinical performance of both treatment options.

This is a non-interventional observational study. Only routine clinical examinations are performed. No additional risks or burdens arise for participants. All measures fall under minimal risk A according to ClinO, Art. 61. Overall risk: Minimal. No invasive procedures or biological sampling. Ethical and legal standards are fully met.

Sex and gender dimensions are not relevant to the topic of the study as the population is determined by patients treated since 2001 and cannot be influenced by the study design.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Patients with at least one extracoronal adhesive attachment for anchoring an RPD and patients with clasp-retained RPD during a 25-year period (2001 - 2025) at the Department for Reconstructive Dentistry or the affiliated student course.
* The attachment or clasp must have been in place for a minimum of six months at the time of clinical follow-up.
* Sufficient availability of medical/dental records
* Age ≥18 years at time of initial treatment.
* Ability to attend a clinical follow-up appointment.

Exclusion Criteria:

* Patients unable to provide informed consent.
* Incomplete or missing documentation of the prosthetic treatment.
* Attachments or clasps inserted less than six months ago.
* Inability to attend the follow-up appointment or language barriers preventing study understanding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective study including all available patients who received an extracoronal adhesive attachment at the University Center for Dental Medicine Basel (UZB) between 2001 and 2025 and a comparable group (same observation group, age and distribution of abutment teeth) with a comparable sample size who received a clasp-retained RPD. Eligible cases will be identified using the relevant billing code entered into the internal billing system
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Patients' satisfaction with extracoronal adhesive attachments (group A) compared to conventional clasp-retained prostheses (group B) on a visual analogue scale (VAS) | From 2001 to present (RDP with retention element has to be in place for at least 6 months)
  The primary objective of this study is to assess patients' satisfaction with extracoronal adhesive attachments (group A) compared to conventional clasp-retained prostheses (group B) on a visual analogue scale (VAS).
  The scale ranges from 0 - 100. A lower score means a worse outcome (satisfaction low) and a higher score a better outcome (satisfaction high). The participants will be instructed and asked to mark a point on the scale according to their satisfaction with the extracoronal adhesive attachment or the clasp-retained prostheses.

SECONDARY OUTCOMES:
Occurrence of biological complications associated with the use of extracoronal adhesive attachments and conventional clasps | From 2001 to present (RDP with retention element has to be in place for at least 6 months)
  At the recall appointment, a clinical examination of the remaining dentition and the prostheses will be performed. The primary assessment will determine whether the abutment tooth with the attachment/clasp remains in situ. The secondary assessment includes a clinical evaluation of the periodontal and endodontic conditions. All biological complications such as caries lesions, tooth fractures, periodontal attachment loss, and endodontic pathologies of the abutment teeth will be reported in a standardized dental record.
  If consent is given, relevant information from the existing dental records will also be extracted for analysis.
Occurrence of technical complications associated with the use of extracoronal adhesive attachments and conventional clasps | From 2001 to present (RDP with retention element has to be in place for at least 6 months)
  At the recall appointment, a clinical examination of the remaining dentition and the prostheses will be performed. The assessment includes a clinical evaluation of the technical condition of the attachment/clasp and the RDP, such as comprise loss of retention between the extracoronal adhesive attachment and the corresponding matrice, loss of the matrice, debonding of the attachment, fracture of the attachment or clasps, deactivation of the clasps, fracture of the removable dental prostheses. The findings will be reported in a standardized dental record.
  If consent is given, relevant information from the dental records will also be extracted for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Zitzmann, Prof. Dr. med. dent. PhD, Study Chair — University of Basel
Locations (1):
- Universitäres Zentrum für Zahnmedizin Basel - Klinik für Rekonstruktive Zahnmedizin, Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
During the clinical visit the questionnaire will be used as a paper case report form. Afterwards the data is transferred to an electronic database for later analysis and in the same step anonymized by using the patients code on the case report for further electronical storage of the collected data. Only study personnel will have access to it. Clinical parameters and patient satisfaction data will be used in encrypted form for statistical evaluation.

REFERENCES:
- [Background] Schaffer H. [Clinical results of partial denture anchorage using extracoronal bonded attachments]. Dtsch Zahnarztl Z. 1990 Jun;45(6):326-8. German. PMID 2269117
- [Background] Besimo C, Gachter M, Jahn M, Hassell T. Clinical performance of resin-bonded fixed partial dentures and extracoronal attachments for removable prostheses. J Prosthet Dent. 1997 Nov;78(5):465-71. doi: 10.1016/s0022-3913(97)70061-1. PMID 9399188
- [Background] Dula LJ, Kelmendi TZ, Shala K, Staka G, Pustina-Krasniqi T, Kosumi S. Attachment-Retained versus Clasp-Retained Removable Partial Dentures: Effects of Retention on Patient Satisfaction. Eur J Dent. 2025 Jul;19(3):823-834. doi: 10.1055/s-0044-1795122. Epub 2024 Dec 30. PMID 39750515
- [Background] Kraljevic I, Glenz F, Jordi C, Zimmermann SD, Joda T, Zitzmann NU. Long-Term Observation of Post Copings Retaining Overdenture Prostheses. Int J Prosthodont. 2020 Mar/Apr;33(2):169-175. doi: 10.11607/ijp.6629. PMID 32069341
- [Background] Zitzmann NU, Rohner U, Weiger R, Krastl G. When to choose which retention element to use for removable dental prostheses. Int J Prosthodont. 2009 Mar-Apr;22(2):161-7. PMID 19418863
- [Background] Brandt S, Winter A, Lauer HC, Romanos G. Retrospective clinical study of 842 clasp-retained removable partial dentures with a metal framework: survival, maintenance needs, and biologic findings. Quintessence Int. 2024 Oct 24;55(9):704-711. doi: 10.3290/j.qi.b5566187. PMID 38985439
- [Background] Garling A, Krummel A, Kern M. Outcomes of resin-bonded attachments for removable dental prostheses. J Prosthodont Res. 2024 Jan 16;68(1):100-104. doi: 10.2186/jpr.JPR_D_22_00306. Epub 2023 May 20. PMID 37211411